CLINICAL TRIAL: NCT01905800
Title: Randomized Multicenter Study of Benign Paroxysmal Positional Vertigo Treatment in Biaxial Rotational Chair
Brief Title: BPPV Treatment in Biaxial Rotational Chair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Camilla Martens, Cand.med, Haukeland University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/980
Record Dates: First submitted 2013-07-15; First posted 2013-07-23 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Benign Paroxysmal Positional Vertigo
Keywords: Vertigo and dizziness.; semicircular canals
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vertigo; Dizziness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Barbecue treatment without acceleration (Active Comparator): Treatment of horizontal BPPV with adapted maneuvers using a biaxial rotational chair and infrared videoscopy goggle. The patient is positioned in supine position and rotated 30 degrees stepwise towards the unaffected ear, thus applying an overall 360 degrees rotation. The patient remains in each position for 30 seconds
  Interventions: Device: Biaxial rotational chair
- Barbecue treatment with acceleartion (Experimental): Treatment of horizontal BPPV with adapted maneuvers using a biaxial rotational chair and infrared videoscopy goggle. The patient starts in supine position and will be rotated about a horizontal axis from head to feet. The patient will be rotated 360 degrees with a succession of eight fast rounds in the axial plane towards the unaffected side.
  Interventions: Device: Biaxial rotational chair
- Placebo treatment (Placebo Comparator): Positional examination of horizontal BPPV with adapted maneuvers using a biaxial rotational chair and infrared videoscopy goggle. The patient is positioned in supine position and rotated 30 degrees stepwise towards the unaffected ear, thus applying a rotation towards the other side.
  Interventions: Device: Biaxial rotational chair

INTERVENTIONS:
Device: Biaxial rotational chair — This chair has a vertical and a horizontal axis of rotation and is lockable in preset positions. It is manually handled and can swivel between two axes in all planes of the semicircular canals for up to 360 degrees or more. Velocity of rotation can be regulated freely.
  Other Names: TRV chair

SUMMARY:
Benign paroxysmal positional vertigo (BPPV) represents the most common cause of labyrinthine vertigo with a lifetime prevalence of 2.4 percent. Onset is most common between the fifth and seventh decades of life. The disease can be a major handicap for the affected patient, and causes a great expense for society. The traditional manual treatment with repositioning maneuvers has greatly improved the possibilities for treatment of BPPV the last decade. However some patients are still difficult to diagnose and treat, and there are some who for health reasons cannot undergo traditional manual treatment. In this perspective there is a demand for a reliable, effective and precise method to treat all semicircular canals for the differentiated patient groups, and the techniques are under continuous development.

DETAILED DESCRIPTION:
There has been extended research to improve the techniques and develop better and more reliable methods for diagnosing and treating BPPV efficiently. An important part in this technique evolution is the development of biaxial rotational chairs that can treat the patients regardless of other health problems.

Mechanical assistance chairs have been designed to diagnose, differentiate and treat more precisely all forms of positional vertigo. The patient is strapped to a chair and fitted with infrared video goggles which identify and quantify the nystagmus in different positions. Dr. John M. Epley developed the Epley Omniax System, an automated, power driven, multi axial patient positioning device that can move the patient into any position to treat the affected canal. This chair is electronically managed. Another mechanical assistance chair, the TRV chair, developed by Thomas Richard-Vitton in Marseille France, became commercially available in 2005. This chair has a vertical and a horizontal axis of rotation and is lockable in preset positions. It is manually handled and can swivel between two axes in all planes of the semicircular canals for up to 360 degrees or more. Velocity of rotation can be regulated freely.

The TRV chair is used by 34 centers worldwide today. Bergen (Norway) was the first place in North-Europe to acquire this chair, and have used it since December 2009. In 2013 Rigshospitalet Denmark started using the TRV chair as well and Oslo University Hospital Rikshospitalet, will have their chair in 2013. The TRV chair opens for treatment that previously was not possible.

The aim of this study is to:

* Evaluate the presence of positional nystagmus in the normal population
* Evaluate the efficacy of D-BBC treatment compared to S-BBC for treatment of lateral canal BPPV in TRV chair
* Examine the serum level of vitamin D in BPPV patients
* Give a detailed description of the method.

ELIGIBILITY:
Inclusion Criteria:

* subjects over 18 years with benign paroxysmal positional vertigo(BPPV)

Exclusion Criteria:

* BPPV previously treated with reposition maneuvers within the last 12 months.
* Cochlear Implant (CI).
* Asymmetrical hearing loss.
* Unusual headache.
* Neurological disease.
* Inner ear disease other than BPPV.
* Semicircular canal paresis.
* Drug that causes dizziness/nystagmus.
* Chemotherapy.
* Hospital admission due to head trauma within the last 12 months.
* Closeness to study group.
* Downbeating nystagmus or upbeating nystagmus without torsional component.
* Extensive spontaneous nystagmus that complicates gait interpretation.
* Cannot tolerate both treatments.
* Pregnancy.
* Bilateral affection of the semicircular canals.
* More than two semicircular canals affected on one side.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-08; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Effect of change in velocity in treatment of lateral canal BPPV | Four years
  Two week cure rate

SECONDARY OUTCOMES:
Effect of change in velocity in treatment of lateral canal BPPV | Four years
  Difference in dynamic barbecue and stepwise barbecue three months after treatment (Cure rate and DHI)

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Martens, MD, Principal Investigator — Haukeland University Hospital; Stein Helge Nordahl Glad, Study Director — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data (IPD) available

REFERENCES:
- [Derived] Martens C, Goplen FK, Aasen T, Gjestad R, Nordfalk KF, Nordahl SHG. Treatment of horizontal canal BPPV-a randomized sham-controlled trial comparing two therapeutic maneuvers of different speeds. Laryngoscope Investig Otolaryngol. 2020 Jun 29;5(4):750-757. doi: 10.1002/lio2.420. eCollection 2020 Aug. PMID 32864448